CLINICAL TRIAL: NCT02335801
Title: The TOSCA Registry: Epidemiology, Clinical and Prognostic Value of Hormonal and Metabolic Deficiencies in Chronic Heart Failure
Brief Title: The TOSCA Registry: Hormonal and Metabolic Deficiencies in Chronic Heart Failure
Acronym: TOSCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Associate Professor, Federico II University
Other Study IDs: TOSCA0001
Record Dates: First submitted 2014-12-09; First posted 2015-01-12 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Chronic Heart Failure
Keywords: heart failure; growth hormone; testosterone; insulin resistance; thyroid hormones; survival
MeSH Terms: conditions — Heart Failure; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples Without DNA — serum for determination of hormonal levels
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to determine whether the presence of metabolic alteration and anabolic deficiencies in patients with chronic heart failure are able to identify a subset of patients with poor outcome.

DETAILED DESCRIPTION:
Despite the effectiveness of the neurohormonal model to explain the progression of heart failure and the many insights that it provided for the development of new therapies, there is increasing clinical evidence that suggests that our current models fail to completely explain the disease progression. Thus, neurohormonal models may be necessary but not sufficient to explain all aspects of disease progression in the failing heart. There is evidence suggesting that in heart failure there is a metabolic imbalance characterized by the predominance of the catabolic status over the anabolic drive.

Aim of this registry is to determine the prevalence of hormone/metabolic deficiencies in heart failure patients and to look for possible association with clinical variables. Moreover, enrolled patients will be followed up for a mean of 2,5 years in order to collect outcome data including all-cause mortality, cardiovascular mortality, hospitalizations.

This is a multi-center observational study involving several Italian Department of Cardiology, Endocrinology, Internal Medicine

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex affected by CHF, secondary to ischemic or idiopathic dilated cardiomyopathy
* left ventricle ejection fraction 40% or less

Exclusion Criteria:

* severe liver disease
* serum creatinine levels >2.5 mg/dl
* history of active cancer with life expectancy below 1 year
* acute coronary syndrome in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with stable chronic heart failure with reduced ejection fraction
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality and hospitalization | every six months (up to 5 years)
  outcome assessed during scheduled visits or phone calls

SECONDARY OUTCOMES:
cardiovascular mortality | every six months (up to 5 years)
  outcome assessed during scheduled visits or phone calls
cardiovascular hospitalizations | every six months (up to 5 years)
  outcome assessed during scheduled visits or phone calls

OTHER OUTCOMES:
reduction in peak oxygen consumption | every six months (up to 5 years)
  outcome assessed during scheduled visits
left ventricular volumes | every six months (up to 5 years)
  outcome assessed during scheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cittadini, Principal Investigator — Federico II University
Locations (17):
- Italy (17):
  - U.O. di Cardiologia 2 IRCCS-Istituto Scientifico di Riabilitazione di Cassano delle Murge, Cassano delle Murge, Bari
  - Santa Maria della Pietà Hospital, Nola, Napoli
  - Policlinico di Bari, Bari
  - Policlinico "Vittorio Emanuele" University of Catania, Catania
  - Unità Operativa di Malattie Cardiovascolari del Policlinico Mater Domini, Catanzaro
  - UOC di Medicina Interna IRCCS Oasi Maria SS, Enna
  - UOC Clinica Medica Dipartimento ad Attività Integrata di Medicina Azienda Ospedaliera-Universitaria S.Anna, Ferrara
  - University of Florence, Florence
  - IRCCS Policlinico San Donato Milanese, Milan
  - Department of Traslational Sciences - Federico II University, Naples
  - AORN V. Monaldi SUN - Centro di diagnosi e cura Cardiomiopatie e Scompenso Cardiaco, Napoli
  - Dipartimento di Scienze Biomediche Avanzate Università degli studi di Napoli Federico II, Napoli
  - U.O.S. Endocrinologia Ospedali Riuniti "Villa Sofia - Cervello", Palermo
  - U.O. di Riabilitazione Cardiologica IRCCS S. Raffaele Pisana, Rome
  - UOC Endocrinologia e Malattie del Metabolismo Policlinico Universitario Gemelli, Rome
  - U.O. di Cardiologia e UTIC Ospedale S. Maria Incoronata dell'Olmo, Salerno
  - Medicina Generale ad Indirizzo Endocrinologico - d.O. Azienda Ospedaliera Universitaria Integrata, Verona

REFERENCES:
- [Background] Cittadini A, Saldamarco L, Marra AM, Arcopinto M, Carlomagno G, Imbriaco M, Del Forno D, Vigorito C, Merola B, Oliviero U, Fazio S, Sacca L. Growth hormone deficiency in patients with chronic heart failure and beneficial effects of its correction. J Clin Endocrinol Metab. 2009 Sep;94(9):3329-36. doi: 10.1210/jc.2009-0533. Epub 2009 Jul 7. PMID 19584187
- [Result] Bossone E, Limongelli G, Malizia G, Ferrara F, Vriz O, Citro R, Marra AM, Arcopinto M, Bobbio E, Sirico D, Caliendo L, Ballotta A, D'Andrea A, Frigiola A, Isgaard J, Sacca L, Antonio C; T.O.S.CA. Investigators. The T.O.S.CA. Project: research, education and care. Monaldi Arch Chest Dis. 2011 Dec;76(4):198-203. doi: 10.4081/monaldi.2011.177. PMID 22567736
- [Result] Arcopinto M, Isgaard J, Marra AM, Formisano P, Bossone E, Vriz O, Vigorito C, Sacca L, Douglas PS, Cittadini A. IGF-1 predicts survival in chronic heart failure. Insights from the T.O.S.CA. (Trattamento Ormonale Nello Scompenso CArdiaco) registry. Int J Cardiol. 2014 Oct 20;176(3):1006-8. doi: 10.1016/j.ijcard.2014.07.003. Epub 2014 Jul 11. No abstract available. PMID 25037691
- [Result] Cittadini A, Marra AM, Arcopinto M, Bobbio E, Salzano A, Sirico D, Napoli R, Colao A, Longobardi S, Baliga RR, Bossone E, Sacca L. Growth hormone replacement delays the progression of chronic heart failure combined with growth hormone deficiency: an extension of a randomized controlled single-blind study. JACC Heart Fail. 2013 Aug;1(4):325-330. doi: 10.1016/j.jchf.2013.04.003. Epub 2013 Aug 5. PMID 24621936
- [Derived] Salzano A, D'Assante R, Iacoviello M, Triggiani V, Rengo G, Cacciatore F, Maiello C, Limongelli G, Masarone D, Sciacqua A, Filardi PP, Mancini A, Volterrani M, Vriz O, Castello R, Passantino A, Campo M, Modesti PA, De Giorgi A, Arcopinto M, Gargiulo P, Perticone M, Colao A, Milano S, Garavaglia A, Napoli R, Suzuki T, Bossone E, Marra AM, Cittadini A; T.O.S.CA. Investigators. Progressive right ventricular dysfunction and exercise impairment in patients with heart failure and diabetes mellitus: insights from the T.O.S.CA. Registry. Cardiovasc Diabetol. 2022 Jun 16;21(1):108. doi: 10.1186/s12933-022-01543-3. PMID 35710369
- [Derived] Cittadini A, Salzano A, Iacoviello M, Triggiani V, Rengo G, Cacciatore F, Maiello C, Limongelli G, Masarone D, Perticone F, Cimellaro A, Perrone Filardi P, Paolillo S, Mancini A, Volterrani M, Vriz O, Castello R, Passantino A, Campo M, Modesti PA, De Giorgi A, Monte IP, Puzzo A, Ballotta A, D'Assante R, Arcopinto M, Gargiulo P, Sciacqua A, Bruzzese D, Colao A, Napoli R, Suzuki T, Eagle KA, Ventura HO, Marra AM, Bossone E; T.O.S.CA. Investigators. Multiple hormonal and metabolic deficiency syndrome predicts outcome in heart failure: the T.O.S.CA. Registry. Eur J Prev Cardiol. 2021 Dec 29;28(15):1691-1700. doi: 10.1093/eurjpc/zwab020. PMID 33693736
- [Derived] Bossone E, Arcopinto M, Iacoviello M, Triggiani V, Cacciatore F, Maiello C, Limongelli G, Masarone D, Perticone F, Sciacqua A, Perrone-Filardi P, Mancini A, Volterrani M, Vriz O, Castello R, Passantino A, Campo M, Modesti PA, De Giorgi A, Monte I, Puzzo A, Ballotta A, Caliendo L, D'Assante R, Marra AM, Salzano A, Suzuki T, Cittadini A; TOSCA Investigators. Multiple hormonal and metabolic deficiency syndrome in chronic heart failure: rationale, design, and demographic characteristics of the T.O.S.CA. Registry. Intern Emerg Med. 2018 Aug;13(5):661-671. doi: 10.1007/s11739-018-1844-8. Epub 2018 Apr 4. PMID 29619769